CLINICAL TRIAL: NCT01355094
Title: Peritoneal Vacuum Therapy to Reduce the Systemic Inflammatory Insult From Intraperitoneal Sepsis/Injury/Hypertension: A Randomized Comparison of Baseline Wall Suction Versus the KCI AbThera™ Abdominal Dressing
Brief Title: Peritoneal Vacuum Therapy to Reduce Inflammatory Response From Abdominal Sepsis/Injury
Acronym: SAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: 3M (Industry); Alberta Health services (Other)
Responsible Party: Principal Investigator, Andrew W Kirkpatrick, Medical Director, Trauma Services, CD, MD, FACS, FRCSC, MHSc, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-23706
Record Dates: First submitted 2011-05-12; First posted 2011-05-17 (Estimated); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Abdominal Compartment Syndrome; Intra-abdominal Hypertension
Keywords: temporary abdomen closure; peritoneal vacuum therapy; open abdomen; abdominal compartment syndrome; intra-abdominal sepsis; intra-abdominal hypertension; critical care
MeSH Terms: conditions — Intra-Abdominal Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- "Stampede" VAC (Active Comparator): Calgary-home-made "Stampede" VAC system with only closed drain bulb suction
  Interventions: Device: "Stampede" VAC
- KCI AbThera (Experimental): commercial AbThera vacuum assisted abdominal closure at 125 mmHg suction
  Interventions: Device: KCI AbThera

INTERVENTIONS:
Device: KCI AbThera — The time that the dressing will be left in place will be left to the discretion of the attending surgeon, but revised practice guidelines mandate either formal abdominal closure or dressing change at 24-96 hours from placement. Upon the first OA dressing change, the surgeon is free to utilize whatever temporary closure they choose.
  Just prior to placement of the dressing, 16 ml (1 table spoon) of blood will be drawn from an existing arterial or venous line (this will qualify as Day 1). The same quantity of blood will be drawn on days 2, 3, 7 and 28 (or hospital discharge, whichever comes first). 15ml of peritoneal fluid will also be collected from the abdomen on the same days or until closure of the abdomen and removal of the dressing.
  Arms: KCI AbThera
Device: "Stampede" VAC — The time that the dressing will be left in place will be left to the discretion of the attending surgeon, but revised practice guidelines mandate either formal abdominal closure or dressing change at 24-96 hours from placement. Upon the first OA dressing change, the surgeon is free to utilize whatever temporary closure they choose.
  Just prior to placement of the dressing, 16 ml (1 table spoon) of blood will be drawn from an existing arterial or venous line (this will qualify as Day 1). The same quantity of blood will be drawn on days 2, 3, 7 and 28 (or hospital discharge, whichever comes first). 15ml of peritoneal fluid will also be collected from the abdomen on the same days or until closure of the abdomen and removal of the dressing.
  Arms: "Stampede" VAC

SUMMARY:
This pilot study will evaluate the effectiveness in actively removing the peritoneal fluid through the use of a commercial suction device compared to passive drainage of the same peritoneal fluid drained through standard surgical drains under bulb suction only, in critically ill patients who require an "open abdomen". Both techniques being used, the commercial KCI AbThera™ device and home made "Stampede" VAC system, are currently approved for use in Canada and used in our facility.

The use or non-use of the open abdomen and its relationship to intra-abdominal hypertension (IAH) and the abdominal compartment syndrome (ACS), the level of IAH must be treated and if so how should be treated - remain controversial. The ultimate treatment for IAH/ACS is to leave the abdominal fascia open after laparotomy, utilizing some form of temporary abdominal closure (TAC) techniques, resulting in an "open abdomen"(OA). The decision to accept an OA can only be made in the operating room and is typically made quite arbitrarily (there is no current standard or protocol),and the TAC used is based on the surgeon's best judgment. The study intends to randomize patients after it has been decided that a TAC is required, which will be applied in the operating room while the patient is fully anesthetized. The only intervention required is to obtain small aliquots (a teaspoonful-15ml) of blood for the evaluation of inflammatory mediators levels, as well as the same volume of intra-peritoneal fluid-that is typically discarded in patients with OA.

DETAILED DESCRIPTION:
Excessive pressure within the peritoneal cavity, known as intra-abdominal hypertension (IAH), can adversely affect not only intra-peritoneal organ function, but also other organ systems throughout the body. When IAH > 20 mmHg induces new organ dysfunction, a potentially lethal condition known as the abdominal compartment syndrome (ACS) is defined. Practically, this syndrome can be considered multi-system organ failure occurring from severe IAH. While the physical effects of IAH/ACS are increasingly being described, the humoral ones, related to IAH-induced ischemia are poorly understood. Recent animal work suggests that aggressively removing intra-peritoneal fluids, assumed to be vasoactive mediator-rich, leads to better systemic outcomes. There is no human data to support this however. Previous attempts at peritoneal drainage in inflammatory conditions such as sepsis and pancreatitis where not conclusive, but this may have been due to the inefficiency of the systems used and the lack of attention to IAH. Recently, efficient systems providing a temporary abdominal closure (TAC) to both drain intra-peritoneal fluids and to control IAH have been introduced. One of these dressing systems, known as the KCI AbThera™ Abdominal Dressing is currently approved for use in Canada as a temporary abdominal closure (TAC) device but its role in ameliorating systemic sepsis/SIRS has not been evaluated.

We propose a randomized trial of using either the "home Calgary Stampede Vac" involving wall suction or the KCI AbThera™ Abdominal Dressing, to dress the abdomen whenever the operative surgeon determines that an open abdomen is warranted to treat the patient.

In general, others have hypothesized that cytokines, especially peritoneal levels, are sensitive indicators of the post-operative inflammatory reaction and may predict complications. In experimental models IL-6 levels are higher in non-survivors. Further, previous work has noted that the blood level of IL-6, which has a longer half life than TNF-α or IL-1β, is a good index of the overall cytokine cascade activation. Thus the main outcomes to be compared will be between mean cytokine levels measured in each of the two treatment groups - to determine if the KCI AbThera™ Abdominal Dressing can significantly reduce the blood concentration of IL-6 when compared with the "Stampede VAC" system. We are hoping to better understand how the body responds to the inflammatory process that naturally occurs during and after an episode of intra-abdominal hypertension, to identify signals or markers of inflammation and infection as well as its progression and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill/injured requiring intensive care unit admission
* Decision regarding the need to utilize an open abdomen technique after the first laparotomy
* Age > 18
* Non-pregnant

Exclusion Criteria:

* Decision to formally close the abdomen after the initial laparotomy
* Patients receiving intra-peritoneal chemotherapy
* Pregnancy
* Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-06; Primary Completion 2022-06 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Systemic inflammatory marker levels and peritoneal fluid inflammatory marker levels | admission to dicharge, expected average of hospital stay 4 weeks.
  Intra-peritoneal and plasma inflammatory mediators will be measured on a treatment allocation basis immediately after initiation of the TAC, and thereafter at 2, 3, 7 and 28 days. The mediators studied will include, but are not limited to TNF-α, IL-1β, IL-6, IL-10, IL-12, and CRP.

SECONDARY OUTCOMES:
Physiological Outcomes | admission to hospital discharge; expected average of hospital stay 4 weeks.
  Determination of the type and activation status of inflammatory cells present in the peritoneal fluid, Measurement of the activation potential of peritoneal fluid, Peritoneal fluid drainage volume, Post-operative fluid balance, Mean 24 hour intra-abdominal pressure (IAP), daily WSACS IAH grading classification, APACHE II score, SOFA score, PaO2/FiO2 ratio, Oxygenation Index, Vasopressor Requirements,RIFLE score, Need for renal replacement therapy, Mean 24 hour lactate level, Mean 24 hour enteral tolerance (if no anastomosis)
Global Outcomes | patients will be followed-up for 6 months
  Death, days with fascial closure for the month after admission, ventilator free days for the month after admission, ICU free days from the month after admission, days free of renal replacement therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W Kirkpatrick, MD, Principal Investigator — Canadian Trauma Trials Collaborative
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Background] Nathens AB, Brenneman FD, Boulanger BR. The abdominal compartment syndrome. Can J Surg. 1997 Aug;40(4):254-8. PMID 9267292
- [Background] Kirkpatrick AW, Baxter KA, Simons RK, Germann E, Lucas CE, Ledgerwood AM. Intra-abdominal complications after surgical repair of small bowel injuries: an international review. J Trauma. 2003 Sep;55(3):399-406. doi: 10.1097/01.TA.0000060248.87046.EE. PMID 14501878
- [Background] Kirkpatrick AW, De Waele JJ, Ball CG, Ranson K, Widder S, Laupland KB. The secondary and recurrent abdominal compartment syndrome. Acta Clin Belg. 2007;62 Suppl 1:60-5. PMID 17469702
- [Background] Ball CG, Kirkpatrick AW, McBeth P. The secondary abdominal compartment syndrome: not just another post-traumatic complication. Can J Surg. 2008 Oct;51(5):399-405. PMID 18841232
- [Background] Ball CG, Kirkpatrick AW. Intra-abdominal hypertension and the abdominal compartment syndrome. Scand J Surg. 2007;96(3):197-204. doi: 10.1177/145749690709600303. No abstract available. PMID 17966744
- [Background] Schein M, Wittmann DH, Aprahamian CC, Condon RE. The abdominal compartment syndrome: the physiological and clinical consequences of elevated intra-abdominal pressure. J Am Coll Surg. 1995 Jun;180(6):745-53. No abstract available. PMID 7773495
- [Background] Balogh ZJ, van Wessem K, Yoshino O, Moore FA. Postinjury abdominal compartment syndrome: are we winning the battle? World J Surg. 2009 Jun;33(6):1134-41. doi: 10.1007/s00268-009-0002-x. PMID 19343417
- [Background] Malbrain ML, Cheatham ML, Kirkpatrick A, Sugrue M, Parr M, De Waele J, Balogh Z, Leppaniemi A, Olvera C, Ivatury R, D'Amours S, Wendon J, Hillman K, Johansson K, Kolkman K, Wilmer A. Results from the International Conference of Experts on Intra-abdominal Hypertension and Abdominal Compartment Syndrome. I. Definitions. Intensive Care Med. 2006 Nov;32(11):1722-32. doi: 10.1007/s00134-006-0349-5. Epub 2006 Sep 12. PMID 16967294
- [Background] Cheatham ML, Malbrain ML, Kirkpatrick A, Sugrue M, Parr M, De Waele J, Balogh Z, Leppaniemi A, Olvera C, Ivatury R, D'Amours S, Wendon J, Hillman K, Wilmer A. Results from the International Conference of Experts on Intra-abdominal Hypertension and Abdominal Compartment Syndrome. II. Recommendations. Intensive Care Med. 2007 Jun;33(6):951-62. doi: 10.1007/s00134-007-0592-4. Epub 2007 Mar 22. PMID 17377769
- [Background] Mayberry JC, Mullins RJ, Crass RA, Trunkey DD. Prevention of abdominal compartment syndrome by absorbable mesh prosthesis closure. Arch Surg. 1997 Sep;132(9):957-61; discussion 961-2. doi: 10.1001/archsurg.1997.01430330023003. PMID 9301607
- [Background] Fietsam R Jr, Villalba M, Glover JL, Clark K. Intra-abdominal compartment syndrome as a complication of ruptured abdominal aortic aneurysm repair. Am Surg. 1989 Jun;55(6):396-402. PMID 2729780
- [Background] Raeburn CD, Moore EE, Biffl WL, Johnson JL, Meldrum DR, Offner PJ, Franciose RJ, Burch JM. The abdominal compartment syndrome is a morbid complication of postinjury damage control surgery. Am J Surg. 2001 Dec;182(6):542-6. doi: 10.1016/s0002-9610(01)00821-2. PMID 11839314
- [Background] Balogh Z, McKinley BA, Cocanour CS, Kozar RA, Holcomb JB, Ware DN, Moore FA. Secondary abdominal compartment syndrome is an elusive early complication of traumatic shock resuscitation. Am J Surg. 2002 Dec;184(6):538-43; discussion 543-4. doi: 10.1016/s0002-9610(02)01050-4. PMID 12488160
- [Background] Ball CG, Kirkpatrick AW, Karmali S, Malbrain ML, Gmora S, Mahabir RC, Doig C, Hameed SM. Tertiary abdominal compartment syndrome in the burn injured patient. J Trauma. 2006 Nov;61(5):1271-3. doi: 10.1097/01.ta.0000198554.25893.f2. No abstract available. PMID 17099543
- [Background] Malbrain ML, Chiumello D, Pelosi P, Bihari D, Innes R, Ranieri VM, Del Turco M, Wilmer A, Brienza N, Malcangi V, Cohen J, Japiassu A, De Keulenaer BL, Daelemans R, Jacquet L, Laterre PF, Frank G, de Souza P, Cesana B, Gattinoni L. Incidence and prognosis of intraabdominal hypertension in a mixed population of critically ill patients: a multiple-center epidemiological study. Crit Care Med. 2005 Feb;33(2):315-22. doi: 10.1097/01.ccm.0000153408.09806.1b. PMID 15699833
- [Background] Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. Crit Care Med. 2001 Jul;29(7):1303-10. doi: 10.1097/00003246-200107000-00002. PMID 11445675
- [Background] Slade E, Tamber PS, Vincent JL. The Surviving Sepsis Campaign: raising awareness to reduce mortality. Crit Care. 2003 Feb;7(1):1-2. doi: 10.1186/cc1876. Epub 2003 Jan 8. PMID 12617727
- [Background] Dellinger RP, Levy MM, Carlet JM, Bion J, Parker MM, Jaeschke R, Reinhart K, Angus DC, Brun-Buisson C, Beale R, Calandra T, Dhainaut JF, Gerlach H, Harvey M, Marini JJ, Marshall J, Ranieri M, Ramsay G, Sevransky J, Thompson BT, Townsend S, Vender JS, Zimmerman JL, Vincent JL; International Surviving Sepsis Campaign Guidelines Committee; American Association of Critical-Care Nurses; American College of Chest Physicians; American College of Emergency Physicians; Canadian Critical Care Society; European Society of Clinical Microbiology and Infectious Diseases; European Society of Intensive Care Medicine; European Respiratory Society; International Sepsis Forum; Japanese Association for Acute Medicine; Japanese Society of Intensive Care Medicine; Society of Critical Care Medicine; Society of Hospital Medicine; Surgical Infection Society; World Federation of Societies of Intensive and Critical Care Medicine. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock: 2008. Crit Care Med. 2008 Jan;36(1):296-327. doi: 10.1097/01.CCM.0000298158.12101.41. PMID 18158437
- [Background] Malbrain ML, Chiumello D, Pelosi P, Wilmer A, Brienza N, Malcangi V, Bihari D, Innes R, Cohen J, Singer P, Japiassu A, Kurtop E, De Keulenaer BL, Daelemans R, Del Turco M, Cosimini P, Ranieri M, Jacquet L, Laterre PF, Gattinoni L. Prevalence of intra-abdominal hypertension in critically ill patients: a multicentre epidemiological study. Intensive Care Med. 2004 May;30(5):822-9. doi: 10.1007/s00134-004-2169-9. Epub 2004 Feb 3. PMID 14758472
- [Background] Regueira T, Hasbun P, Rebolledo R, Galindo J, Aguirre M, Romero C, Castillo L, Bugedo G, Hernandez G. Intraabdominal hypertension in patients with septic shock. Am Surg. 2007 Sep;73(9):865-70. PMID 17939414
- [Background] Chow AW, Evans GA, Nathens AB, Ball CG, Hansen G, Harding GK, Kirkpatrick AW, Weiss K, Zhanel GG. Canadian practice guidelines for surgical intra-abdominal infections. Can J Infect Dis Med Microbiol. 2010 Spring;21(1):11-37. doi: 10.1155/2010/580340. No abstract available. PMID 21358883
- [Background] Marshall JC, Innes M. Intensive care unit management of intra-abdominal infection. Crit Care Med. 2003 Aug;31(8):2228-37. doi: 10.1097/01.CCM.0000087326.59341.51. PMID 12973184
- [Background] Goins WA, Rodriguez A, Joshi M, Jacobs D. Intra-abdominal abscess after blunt abdominal trauma. Ann Surg. 1990 Jul;212(1):60-5. doi: 10.1097/00000658-199007000-00009. PMID 2363605
- [Background] Landow L, Andersen LW. Splanchnic ischaemia and its role in multiple organ failure. Acta Anaesthesiol Scand. 1994 Oct;38(7):626-39. doi: 10.1111/j.1399-6576.1994.tb03969.x. PMID 7839769
- [Background] Welborn MB, Oldenburg HS, Hess PJ, Huber TS, Martin TD, Rauwerda JA, Wesdorp RI, Espat NJ, Copeland EM 3rd, Moldawer LL, Seeger JM. The relationship between visceral ischemia, proinflammatory cytokines, and organ injury in patients undergoing thoracoabdominal aortic aneurysm repair. Crit Care Med. 2000 Sep;28(9):3191-7. doi: 10.1097/00003246-200009000-00013. PMID 11008981
- [Background] Ivatury RR, Porter JM, Simon RJ, Islam S, John R, Stahl WM. Intra-abdominal hypertension after life-threatening penetrating abdominal trauma: prophylaxis, incidence, and clinical relevance to gastric mucosal pH and abdominal compartment syndrome. J Trauma. 1998 Jun;44(6):1016-21; discussion 1021-3. doi: 10.1097/00005373-199806000-00014. PMID 9637157
- [Background] Fink MP, Delude RL. Epithelial barrier dysfunction: a unifying theme to explain the pathogenesis of multiple organ dysfunction at the cellular level. Crit Care Clin. 2005 Apr;21(2):177-96. doi: 10.1016/j.ccc.2005.01.005. PMID 15781156
- [Background] Rongione AJ, Kusske AM, Ashley SW, Reber HA, McFadden DW. Interleukin-10 prevents early cytokine release in severe intraabdominal infection and sepsis. J Surg Res. 1997 Jul 1;70(2):107-12. doi: 10.1006/jsre.1997.5071. PMID 9237883
- [Background] Yao YM, Redl H, Bahrami S, Schlag G. The inflammatory basis of trauma/shock-associated multiple organ failure. Inflamm Res. 1998 May;47(5):201-10. doi: 10.1007/s000110050318. PMID 9657252
- [Background] Wortel CH, van Deventer SJ, Aarden LA, Lygidakis NJ, Buller HR, Hoek FJ, Horikx J, ten Cate JW. Interleukin-6 mediates host defense responses induced by abdominal surgery. Surgery. 1993 Sep;114(3):564-70. PMID 7690162
- [Background] Scheingraber S, Bauerfeind F, Bohme J, Dralle H. Limits of peritoneal cytokine measurements during abdominal lavage treatment for intraabdominal sepsis. Am J Surg. 2001 Apr;181(4):301-8. doi: 10.1016/s0002-9610(01)00587-6. PMID 11438263
- [Background] van Berge Henegouwen MI, van der Poll T, van Deventer SJ, Gouma DJ. Peritoneal cytokine release after elective gastrointestinal surgery and postoperative complications. Am J Surg. 1998 Apr;175(4):311-6. doi: 10.1016/s0002-9610(98)00010-5. PMID 9568659
- [Background] Jansson K, Redler B, Truedsson L, Magnuson A, Matthiessen P, Andersson M, Norgren L. Intraperitoneal cytokine response after major surgery: higher postoperative intraperitoneal versus systemic cytokine levels suggest the gastrointestinal tract as the major source of the postoperative inflammatory reaction. Am J Surg. 2004 Mar;187(3):372-7. doi: 10.1016/j.amjsurg.2003.12.019. PMID 15006565
- [Background] Hendriks T, Bleichrodt RP, Lomme RM, De Man BM, van Goor H, Buyne OR. Peritoneal cytokines predict mortality after surgical treatment of secondary peritonitis in the rat. J Am Coll Surg. 2010 Aug;211(2):263-70. doi: 10.1016/j.jamcollsurg.2010.03.038. Epub 2010 Jun 26. PMID 20670866
- [Background] Holzheimer RG, Schein M, Wittmann DH. Inflammatory response in peritoneal exudate and plasma of patients undergoing planned relaparotomy for severe secondary peritonitis. Arch Surg. 1995 Dec;130(12):1314-9; discussion 1319-20. doi: 10.1001/archsurg.1995.01430120068010. PMID 7492280
- [Background] Martineau L, Shek PN. Peritoneal cytokine concentrations and survival outcome in an experimental bacterial infusion model of peritonitis. Crit Care Med. 2000 Mar;28(3):788-94. doi: 10.1097/00003246-200003000-00030. PMID 10752831
- [Background] Antonelli M, Fumagalli R, Cruz DN, Brienza N, Giunta F. PMX endotoxin removal in the clinical practice: results from the EUPHAS trial. Contrib Nephrol. 2010;167:83-90. doi: 10.1159/000315922. Epub 2010 Jun 1. PMID 20519902
- [Background] Nakamura M, Oda S, Sadahiro T, Hirayama Y, Watanabe E, Tateishi Y, Nakada TA, Hirasawa H. Treatment of severe sepsis and septic shock by CHDF using a PMMA membrane hemofilter as a cytokine modulator. Contrib Nephrol. 2010;166:73-82. doi: 10.1159/000314855. Epub 2010 May 7. PMID 20472994
- [Background] Ratanarat R, Brendolan A, Piccinni P, Dan M, Salvatori G, Ricci Z, Ronco C. Pulse high-volume haemofiltration for treatment of severe sepsis: effects on hemodynamics and survival. Crit Care. 2005 Aug;9(4):R294-302. doi: 10.1186/cc3529. Epub 2005 Apr 28. PMID 16137340
- [Background] Caronna R, Benedetti M, Morelli A, Rocco M, Diana L, Prezioso G, Cardi M, Schiratti M, Martino G, Fanello G, Papini F, Farelli F, Meniconi RL, Marengo M, Dinatale G, Chirletti P. Clinical effects of laparotomy with perioperative continuous peritoneal lavage and postoperative hemofiltration in patients with severe acute pancreatitis. World J Emerg Surg. 2009 Dec 16;4:45. doi: 10.1186/1749-7922-4-45. PMID 20015376
- [Background] Silva E, de Figueiredo LF, Colombari F. Prowess-shock trial: a protocol overview and perspectives. Shock. 2010 Sep;34 Suppl 1:48-53. doi: 10.1097/SHK.0b013e3181e7e97b. PMID 20523271
- [Background] Jennings WC, Wood CD, Guernsey JM. Continuous postoperative lavage in the treatment of peritoneal sepsis. Dis Colon Rectum. 1982 Oct;25(7):641-3. doi: 10.1007/BF02629531. PMID 7128362
- [Background] De Waele JJ, Hesse UJ, Pattyn P, Decruyenaere J, de Hemptinne B. Postoperative lavage and on demand surgical intervention in the treatment of acute necrotizing pancreatitis. Acta Chir Belg. 2000 Feb;100(1):16-20. PMID 10776522
- [Background] Schwarz A, Bolke E, Peiper M, Schulte am Esch J, Steinbach G, van Griensven M, Orth K. Inflammatory peritoneal reaction after perforated appendicitis: continuous peritoneal lavage versus non lavage. Eur J Med Res. 2007 May 29;12(5):200-5. PMID 17513191
- [Background] Buanes TA, Andersen GP, Jacobsen U, Nygaard K. Perforated appendicitis with generalized peritonitis. Prospective, randomized evaluation of closed postoperative peritoneal lavage. Eur J Surg. 1991 Apr;157(4):277-9. PMID 1677283
- [Derived] Bjorck M, Kirkpatrick AW, Cheatham M, Kaplan M, Leppaniemi A, De Waele JJ. Amended Classification of the Open Abdomen. Scand J Surg. 2016 Mar;105(1):5-10. doi: 10.1177/1457496916631853. Epub 2016 Feb 29. PMID 26929286
- [Derived] Kirkpatrick AW, Roberts DJ, Faris PD, Ball CG, Kubes P, Tiruta C, Xiao Z, Holodinsky JK, McBeth PB, Doig CJ, Jenne CN. Active Negative Pressure Peritoneal Therapy After Abbreviated Laparotomy: The Intraperitoneal Vacuum Randomized Controlled Trial. Ann Surg. 2015 Jul;262(1):38-46. doi: 10.1097/SLA.0000000000001095. PMID 25536308
- [Derived] Roberts DJ, Jenne CN, Ball CG, Tiruta C, Leger C, Xiao Z, Faris PD, McBeth PB, Doig CJ, Skinner CR, Ruddell SG, Kubes P, Kirkpatrick AW. Efficacy and safety of active negative pressure peritoneal therapy for reducing the systemic inflammatory response after damage control laparotomy (the Intra-peritoneal Vacuum Trial): study protocol for a randomized controlled trial. Trials. 2013 May 16;14:141. doi: 10.1186/1745-6215-14-141. PMID 23680127